CLINICAL TRIAL: NCT01910103
Title: Comparison of Diagnostic Performance of Digital Breast Tomosynthesis and Ultrasound in Women With Dense Breasts
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung Min Chang, Clinical Assistant Professor, Seoul National University Hospital
Other Study IDs: D-1303-051-472
Record Dates: First submitted 2013-06-24; First posted 2013-07-29 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Breast Neoplasms
Keywords: Breast Neoplasms/radiography; Mammography/methods; Mass Screening; Tomography, X-Ray Computed/methods; Predictive Value of Tests; False Positive Reactions
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Diagnostic performance of digital breast tomosynthesis (DBT) would be not inferior to the that of breast ultrasound in women with dense breast.

DETAILED DESCRIPTION:
1. Patients with dense breast will be examined for the detection of breast cancer by imaging studies.
2. The imaging including digital breast tomosynthesis (DBT), physician-performed bilateral whole breast ultrasonography will be performed according to a standard protocol.Interpretation will be conducted independently and classified according to the Breast Imaging Reporting and Data System (BI-RADS) by experienced radiologists.
3. Definitive information about the presence of malignancy will be obtained by biopsy directed by the imaging method best depicting the lesion with 14-g or 11-g needle devices or needle localized excision. The absence of breast cancer was determined by means of biopsy, the absence of positive findings on repeat imaging and clinical examination, or both at follow-up.
4. The diagnostic yield of digital breast tomosynthesis (DBT) compared to ultrasonography will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Women aged at 20 years
* Women who had heterogeneously dense or extremely dense parenchyma, either by prior mammography report or by review of prior mammograms
* Signed study-specific informed consent prior to registration

Exclusion Criteria:

* Had breast surgery
* Had breast core biopsy performed within the prior 6 months on the study

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women undergoing mammography and breast US for screening or diagnostic purpose
Sampling Method: Non-Probability Sample
Enrollment: 825 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance (AUC: area of under ROC curve) of DBT and US | one year
  The primary endpoint will be an analysis of the diagnostic performance of DBT to that of US for detecting breast cancer in the screening and diagnostic setting. The hypothesis is that DBT is not inferior to US for detecting breast cancer.

SECONDARY OUTCOMES:
Diagnostic sensitivity, sensitivity, negative predictive value, and positive predictive value of DBT and US for detecting breast cancer. | One year
  We will calculate diagnostic sensitivity (%), sensitivity (%), negative predictive value (%), and positive predictive alue (%) of the DBT and US for the detection of breast cancer on a per-patient basis by using a BI-RADS score of 4 or 5 considered as test-positive and a BI-RADS score of 1, 2, or 3 considered as test-negative.
  Cases of women undergoing biopsy with malignant disease results were considered disease-positive. Cases of women with concordant benign biopsy results and women not undergoing biopsy with no evidence of breast malignancy after 1 year of clinical follow-up were considered diase-negative.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Min Chang, M.D., Ph.D., Principal Investigator — Department of Radiology, Seoul National University Hospital
Locations (1):
- Department of Radiology, Seoul National University Hospital, Seoul, South Korea